CLINICAL TRIAL: NCT00123175
Title: Levonorgestrel Containing Intrauterine Device in the Treatment of Endometrial Hyperplasia Without Atypia
Brief Title: Treatment of Endometrial Hyperplasia With an Intrauterine Device (IUD)
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study has never received funding and has never been initiated
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: Center for Research on Women and Newborn Health (Unknown)
Responsible Party: Principal Investigator, Richard S. Legro, M.D., Professor, Obstetrics and Gynecology and Public Health Sciences, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 21012
Record Dates: First submitted 2005-07-20; First posted 2005-07-22 (Estimated); Last update posted 2013-01-08 (Estimated); Status verified 2013-01

CONDITIONS: Endometrial Hyperplasia
Keywords: Endometrial Hyperplasia without atypia
MeSH Terms: conditions — Endometrial Hyperplasia | interventions — Intrauterine Devices

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Intrauterine Device — Mirena and Provera
  Other Names: Medroxyprogesterone Acetate and Progestins

SUMMARY:
The purpose of this research is to determine the effectiveness of the intrauterine device (IUD) called Mirena when compared to the Provera tablets used in treating this condition.

DETAILED DESCRIPTION:
Endometrial hyperplasia without atypia is a condition usually caused by excessive stimulation of the uterine lining (endometrium) by estrogens, and may cause irregular bleeding as a presenting symptom, but rarely may progress to endometrial cancer, which makes treatment important. The only treatment approved so far is medroxyprogesterone acetate tablets (progesterone), also known as Provera.

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis of simple or complex endometrial hyperplasia without atypia
* Normal pap smear within one year

Exclusion Criteria:

* Diabetes
* Family history of endometrial cancer
* Contraindications for the intrauterine device

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-09; Primary Completion 2011-09 (Estimated); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
Pathologic examination of the specimens obtained by endometrial biopsy to determine the regression of endometrial hyperplasia without atypia compared to Provera | 90 days

SECONDARY OUTCOMES:
Side effects | 90 days
Bleeding profile | 90 days
Estradiol and progesterone levels | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Richard Legro, M.D., Principal Investigator — Penn State University College of Medicine